CLINICAL TRIAL: NCT05189158
Title: Ventilatory Responses to Hypercapnic and Hypoxic Conditions in Hyperventilants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B076201836758 -2
Record Dates: First submitted 2021-10-18; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Hyperventilation Syndrome; Hypercapnia; Hypoxia
MeSH Terms: conditions — Hypercapnia; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HVS- (Other): subjects with no complaint AND a Nijmegen questionnaire score of < 23/64 AND a negative hyperventilation provocation test (criteria revised in 2021) (HVS-)
  Interventions: Diagnostic Test: Hypercapnic hyperoxic ventilatory response; Diagnostic Test: Hypoxic eucapnic ventilatory response
- HVS+ (Other): subjects with complaints AND a Nijmegen questionnaire score of ≥23/64 AND a negative hyperventilation provocation test (criteria revised in 2021) (HVS+)
  Interventions: Diagnostic Test: Hypercapnic hyperoxic ventilatory response; Diagnostic Test: Hypoxic eucapnic ventilatory response

INTERVENTIONS:
Diagnostic Test: Hypercapnic hyperoxic ventilatory response — The hypercapnic ventilatory response (HCVR) described by Read in 1967 (Read's rebreathing method) is a clinical way to assess the central and peripheric sensitivity to CO2, using a small bag (4-6 l) to achieve prompt equilibrium between the apparatus compartments and the lungs.
  By rebreathing a hyperoxic mixture with an initial composition of 70% O2, 7% CO2 and 23% N2, this equilibrium is assumed to be achieved after 15 seconds of rebreathing, when the relationship between VE and PetCO2 has become linear.
Diagnostic Test: Hypoxic eucapnic ventilatory response — The hypoxic eucapnic ventilatory response (HOVR) is a clinical way to assess the peripheric chemosensitivity to O2, using a small bag (4-6 l) to rebreathe a gas mixture initially composed of 20% O2, 0% CO2 and Δ% N2. Eucapnia is achieved by the activation of a CO2 reabsorption cell during the course of the test.

SUMMARY:
For almost a century, many hypotheses have converged on the idea of altered chemosensitivity in patients suffering from hyperventilation syndrome (HVS).

Given the evolution of current technical equipment and the ability to maximise true positives in HVS ( using the revised hyperventilation provocation test), it seems reasonable to investigate central and peripheral chemosensitivities in HVS subjects.

DETAILED DESCRIPTION:
In the inter-war period, many medical investigators who studied the hyperventilation syndrome (HVS) had already questioned the chemosensitivity to CO2 in HVS patients, without being able to explore it for all intents and purposes.

It was subsequently observed that although HVS is not systematically linked to manifest resting hypocapnia, it is nevertheless systematically correlated with significant variability and complexity of ventilation.

This is consistent with the observations of an increased plant gain in HVS, to be related to an increased loop gain (due to instability of controller gain feedback).

On the other hand, some authors already noted that, when capnia is chronically compromised in HVS, it can be greatly altered by small, transient and barely perceptible increases in VE: a 10% increase in VE could indeed halve PetCO2, while a sigh would be able to decrease PetCO2 by up to 15mmHg.

More recently, teh assumption was made that peripheral chemosensitivity may be impaired in HVS patients.

For all these considerations, it seems reasonable to investigate central and peripheral chemosensitivities in identified HVS subjects on the basis of an objective test, such as the induced hyperventilation test.

ELIGIBILITY:
Inclusion Criteria:

* A plethysmography within subject's predicted values
* A negative metacholine test (no documented allergy)
* A hyperventilation provocation test result that is consistent with the Nijmegen questionnaire score, confirming either group classification (HVS+ or HVS-)

Exclusion Criteria:

* Each of the following known or documented conditions: chronic bronchitis (COPD), emphysema, asthma, cardiac disorder, neurological disorder, gastrointestinal disorder, thyroid disorder or psychological/psychiatric disorder
* Suspicious cardio-pulmonary exercise testing (CPET) with cardiac or respiratory limitation
* Pregnant women or women in the process of becoming pregnant
* Persons with a diving practice (amateur or professional),
* High-level athletes,
* Active smokers and
* persons using morphine, and/or barbiturates, and/or anxiolytics and/or sleeping pills

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
The slope of the ventilatory response to hypercapnia (HCVR) | baseline - during the test
  Ventilation increase (litres/min) per unit increase in PetCO2 (mmHg) using Read's method
The slope of the ventilatory response to hypoxia (HOVR) | baseline - during the test
  Ventilation increase (litres/min) per unit decrease in SpO2 (%) using Read's method
Ventilatory recruitment threshold (VRT) of the HCVR | baseline - during the test
  From the average baseline ventilation and PetCO2, the VRT id the PetCO2 level at which the ventilatory response is activated
Ventilatory recruitment threshold (VRT) of the HOVR | baseline - during the test
  From the average baseline ventilation and SpO2, the VRT is the level of SpO2 at which the ventilatory response is activated

SECONDARY OUTCOMES:
Extrapolated apnoeic threshold of the HCVR | baseline - during the test
  PetCO2 level above which apnoea (zero ventilation) is disrupted, obtained from the extrapolation of the HCVR at the X-axis intersection (when VE=0 l/min)
Dyspnea | baseline, end of the test
  Visual analogic scale (VAS) of dyspnea, from 0 (no dyspnea) to 10 (maximal dyspnea)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU St Pierre, Brussels, Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No